CLINICAL TRIAL: NCT00004125
Title: A Phase III Study of Doxorubicin-Cyclophosphamide Therapy Followed by Paclitaxel or Docetaxel Given Weekly or Every 3 Weeks in Patients With Axillary Node-Positive Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Stage II or Stage IIIA Breast Cancer That Has Spread to the Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067353; E1199; CLB-49906; NCCTG-E1199; SWOG-E1199
Record Dates: First submitted 1999-12-10; First posted 2003-08-25 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Paclitaxel; Tamoxifen; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Drug: tamoxifen citrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of chemotherapy is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of combination chemotherapy in treating women who have stage II or stage IIIA breast cancer that has spread to the lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival and overall survival in patients with node-positive or high-risk node-negative operable stage II or IIIA breast cancer treated with docetaxel or paclitaxel after doxorubicin and cyclophosphamide.
* Determine whether the weekly administration of paclitaxel or docetaxel for 12 weeks improves disease-free survival and overall survival when compared with the conventional schedule of every 3 weeks for 4 courses after doxorubicin and cyclophosphamide in this patient population.
* Compare the toxic effects of docetaxel and paclitaxel when administered weekly for 12 weeks versus every 3 weeks for 4 courses in these patients.
* Compare the toxicity of paclitaxel administered every 3 weeks for 4 courses or weekly for 12 weeks to that of docetaxel administered on the same schedules in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to estrogen receptor status (positive vs negative vs unknown), nodal status (0 positive nodes vs 1-3 positive nodes vs 4-9 positive nodes vs at least 10 positive nodes), tumor size (no more than 5 cm vs more than 5 cm vs unknown), and type of prior surgery (mastectomy vs breast conservation surgery). Patients are randomized to one of four treatment arms.

* Arm I: Patients receive doxorubicin IV and cyclophosphamide IV every 3 weeks for 4 courses (weeks 1-12). Beginning at week 13, patients receive paclitaxel IV over 3 hours every 3 weeks for 4 courses.
* Arm II: Patients receive doxorubicin and cyclophosphamide as in arm I. Beginning at week 13, patients receive paclitaxel IV over 1 hour weekly for 12 weeks.
* Arm III: Patients receive doxorubicin and cyclophosphamide as in arm I. Beginning at week 13, patients receive docetaxel IV over 1 hour every 3 weeks for 4 courses.
* Arm IV: Patients receive doxorubicin and cyclophosphamide as in arm I. Beginning at week 13, patients receive docetaxel IV over 1 hour weekly for 12 weeks.

Within 4 weeks after completion of chemotherapy, patients with estrogen and/or progesterone receptor positive tumors receive oral tamoxifen daily for 5 years.

After completion of all chemotherapy, patients with prior segmental mastectomy receive radiotherapy once daily 5 days per week for 5-6 weeks. Patients with prior modified radical mastectomy may receive radiotherapy after chemotherapy completion at the investigator's discretion.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 5,000 patients will be accrued for this study within 1.27 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed operable stage IIA, IIB, or IIIA adenocarcinoma of the breast with histologically involved lymph nodes (T1, 2, or 3; N1 or 2; M0) OR high-risk node-negative disease (T2 or 3; N0)

  * Primary tumor at least 2.1 cm in diameter for node-negative disease
  * Bilateral breast disease allowed if at least 1 primary tumor meets the criteria above
* Must have had at least 6 axillary lymph nodes removed at dissection and at least one node positive for metastasis OR
* Sentinel node biopsy negative for metastasis (sentinel node biopsy positive allowed if enrolled on American College of Surgery Trial Z0011 and have beenrandomized to receive no axillary dissection)

  * Additional axillary nodes may be obtained provided they are also negative for metastasis
* Complete tumor removal by either a modified radical mastectomy or local excision plus axillary lymph node dissection (i.e., breast conservation therapy) or sentinel node biopsy

  * Tumor-free margins at least 1 mm for both invasive and noninvasive carcinoma except for lobular carcinoma in situ (less than 1 mm allowed)
* Concurrent enrollment on American College of Surgery Trial Z0010, Z0011, or NSABP B-32 allowed
* Hormone receptor status:

  * Estrogen receptor status positive, negative, or unknown

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No history of myocardial infarction
* No congestive heart failure
* No significant ischemic or valvular heart disease

Other:

* No other prior invasive malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No hypersensitivity to paclitaxel or docetaxel or other similarly formulated drugs (with Cremophor or polysorbate)
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for breast cancer

Endocrine therapy:

* Prior tamoxifen of no more than 4 weeks duration for breast cancer allowed
* Prior tamoxifen or other selective estrogen receptor modulator (SERM) for chemoprevention (e.g., Breast Cancer Prevention Trial) or for other indications (e.g., osteoporosis) allowed
* No concurrent tamoxifen or other SERMs

Radiotherapy:

* No prior radiotherapy for this malignancy
* At least 2 weeks since prior radiotherapy to the breast for ductal carcinoma in situ

Surgery:

* See Disease Characteristics
* Less than 84 days since prior surgical procedure to adequately treat primary tumor

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11-16 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Sparano, MD, Study Chair — Albert Einstein College of Medicine; Edith A. Perez, MD, Study Chair — Mayo Clinic; Silvana Martino, DO, Study Chair — Saint John's Cancer Institute; Vicky E. Jones, MD, Study Chair — University of California, San Diego
Locations (48):
- United States (48):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Sparano JA, Wang M, Martino S, Jones V, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Weekly paclitaxel in the adjuvant treatment of breast cancer. N Engl J Med. 2008 Apr 17;358(16):1663-71. doi: 10.1056/NEJMoa0707056. PMID 18420499
- [Result] Sparano JA, Wang M, Martino S, et al.: Phase III study of doxorubicin-cyclophosphamide followed by paclitaxel or docetaxel given every 3 weeks or weekly in patients with axillary node-positive or high-risk node-negative breast cancer: results of North American Breast Cancer Intergroup Trial E1199. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-48, 2005.
- [Derived] Sparano JA, Zhao F, Martino S, Ligibel JA, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Long-Term Follow-Up of the E1199 Phase III Trial Evaluating the Role of Taxane and Schedule in Operable Breast Cancer. J Clin Oncol. 2015 Jul 20;33(21):2353-60. doi: 10.1200/JCO.2015.60.9271. Epub 2015 Jun 15. PMID 26077235